CLINICAL TRIAL: NCT00353990
Title: Bioavailability, Pharmacokinetics and Pharmacodynamics of Insulin Aspart Administered in the Duodenum in Healthy Volunteers - an Open Single Blinded and Uncontrolled Explorative Trial
Brief Title: Bioavailability of Insulin Administered in Duodenum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-002803-15
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus
Keywords: insulin; bioavailability; duodenum; infusion; healthy; diabetes; absorption
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin Aspart

SUMMARY:
A study of the bioavailability of insulin after infusion in the duodenum in healthy volunteers.

DETAILED DESCRIPTION:
METHODOLOGY All subjects will be admitted fasting to the Clinical Trial Unit at Århus Community Hospital at 8 a.m. A Gastrointestinal tube will be placed in Duodenum distal to papilla Vaterii with a pH of approximately 7.0 as measured by the pH meter distal in the tube. An indwelling catheter for glucose infusion (20 %) in cases of hypoglycaemia will be placed in an antecubital vein. In the contralateral anticubital vein a catheter will be placed for blood sampling. All subjects will have 4 tests with duodenal infusion of the insulin Aspart solution. The first 4 volunteers will receive 4 doses of insulin Aspart solution in 1 ml (150, 300, 600 and 1000 IU) with 3-6 hours apart. Blood sampling for Insulin Aspart, total insulin, and glucose (Beckmann apparatus) will be done every 10 minutes the first two hours, and then every 20 minutes. When final the subjects will receive a meal before leaving the hospital.

Based on data from the pilot a dose will be determined for the remaining 8 subjects. These will then based again on results from the pilot on two separate study days receive 4 infusions with 3-6 hours split. Two infusions will be at pH 7 and two infusions will be more proximal at a pH of 5.5 (two different insulin concentrations but the same dose given at the two places in Duodenum). Frequency and interval of blood sampling in the second part will be determined by results from the pilot study. For comparison with the clinical situation and estimation of bioavailability all subjects will receive a subcutaneous and an intravenous (iv) bolus injection of 6 IU of insulin Aspart. The iv injection will be followed by blood sampling for three hours as above, but every 5 minutes the first two hours, and the sc injection will be followed by blood sampling for three hours as above, but again with 10 minutes interval the first two hours.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy Volunteers
* Age >18 - < 50 years
* BMI 18-30 kg/m2

Exclusion Criteria:

* Any history of gastrointestinal or endocrine disorders (e.g. diabetes mellitus)
* pregnancy or nursing
* suspected or known allergy towards the drug
* Participation in other research trials within 3 months before the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To define the bioavailability of a solution of insulin Aspart infused in the Duodenum

SECONDARY OUTCOMES:
Evaluate pharmacokinetics of insulin following duodenal administration
Evaluate intra- and intersubjects variation in pharmacokinetic
Evaluate pharmacodynamics of insulin
To assess any safety issues
Explore any influence of PH/ insulin concentration on PK /PD parameters

CONTACTS AND LOCATIONS:
Overall Officials: Torben Laursen, MD, DMSc, Ph.D., Principal Investigator — Department of Clinical Pharmacology, Aarhus Sygehus; Charlotte A Ihlo, MD, Principal Investigator — Department of Endocrinilogy, Universityhospital of Aarhus
Locations (1):
- Medical Department M, Aarhus, Aarhus, Denmark